CLINICAL TRIAL: NCT01682577
Title: Bioequivalence Study of 4 mg Perindopril Tablets Produced by PT Dexa Medica in Comparison With the Reference Tablets (Prexum® 4 mg, Servier)Under Fasting Condition
Brief Title: Bioequivalence Study of Two Formulations of Perindopril 4 mg Tablet Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PR.122/EQL/2008
Record Dates: First submitted 2012-09-03; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Perindopril; Perindoprilat; Bioequivalence; Pharmacokinetic; Angiotensin-converting enzyme inhibitor
MeSH Terms: interventions — Perindopril

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perindopril 4 mg tablets of PT Dexa Medica (Experimental): Group I (Test product): each tablet contains perindopril tert-butylamine salt 4 mg.
  A single dose of perindopril tablet of PT Dexa Medica was given to each of study subjects.
  Interventions: Drug: Perindopril 4 mg tablets of PT Dexa Medica
- Perindopril 4 mg tablets of Servier (Active Comparator): Group II (Reference product) : each tablet contains perindopril tert-butylamine salt 4 mg.
  A single dose of perindopril (Prexum) tablets of Servier was given to each of study subjects.
  Interventions: Drug: Perindopril 4 mg tablets of Servier

INTERVENTIONS:
Drug: Perindopril 4 mg tablets of PT Dexa Medica — Test product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Test Product: Perindopril 4 mg tablets of PT Dexa Medica.; Each tablet contains perindopril tert-butylamine salt 4 mg
  Arms: Perindopril 4 mg tablets of PT Dexa Medica
Drug: Perindopril 4 mg tablets of Servier — Reference product was given as a single dose, under the procedure as described in the Section: Detailed description of the study.
  Other Names: Reference product: Prexum® 4 mg, produced by Servier.; Each tablet contains Perindopril tert-butylamine salt 4 mg.
  Arms: Perindopril 4 mg tablets of Servier

SUMMARY:
The objective of this study was to find out whether the bioavailability of PT Dexa Medica's formulation of 4 mg perindopril tert-butylamine tablets was equivalent to that of the innovator's product (Prexum® 4 mg, Servier).

DETAILED DESCRIPTION:
The participating subjects were required to have an overnight fast and in the next morning were given orally one tablet of the test drug (Perindopril 4 mg tablets of PT Dexa Medica) or one tablet of the reference drug (Prexum® 4 mg, Servier).

Blood samples were drawn immediately before taking the drug (control), and at 20, 40 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 192 hours after drug administration.

Three weeks after the first drug administration (washout period), the procedure was repeated using the alternate drug.

The pharmacokinetic parameters, including AUCt, AUCinf, Cmax, t max, and t1/2, were determined based on the concentrations of the perindopril parent compound and the metabolite perindoprilat, using high-performance liquid chromatography method with tandem mass spectrometry detector (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Aged 18-55 years inclusive
* A body mass index in the range of 18-25 kg/m2
* Able to participate, communicate well with the investigators and willing to give informed consent
* Non-smokers
* Vital signs (after 10 minutes resting) are within the following ranges:

  * systolic blood pressure 100-125 mmHg
  * diastolic blood pressure 60-80 mmHg
  * pulse rate 60-90 bpm

Exclusion Criteria:

* Pregnant or lactating women
* Known hypersensitivity or contraindication to perindopril
* Intake of any prescription drug within 14 days of this study's first dosing day
* Intake of any non-prescription drug, food supplement, or herbal medicine within 7 days of this study's first dosing day
* History or presence of any liver dysfunction (ALT, alkaline phosphatase, total bilirubin ≥ 1.5 ULN)
* History of any bleeding or coagulation disorders
* Clinically significant ECG abnormalities
* Clinically significant haematology abnormalities
* Renal insufficiency (plasma creatinine concentration ≥ 1.4 mg/dL)
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drug
* A donation or loss of 500 mL (or more) of blood within 3 months before this study's first dosing day
* A positive hepatitis B surface antigen (HBsAg), anti-HCV, and anti-HIV
* History of drug or alcohol abuse within 12 months prior to screening of this study
* Participation in a previous study within 3 months of this study's first dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve (AUC)of perindopril parent compound | 192 hours
  Relative bioavailability (primarily measured by AUCt and AUCinf) between two perindopril 4 mg tablet formulations (test and reference formulations) under fasting condition. The AUC was measured based on the plasma concentration of perindopril parent compound.
Area under concentration-time curve (AUC)of perindoprilat | 192 hours
  Relative bioavailability (primarily measured by AUCt and AUCinf) between two perindopril 4 mg tablet formulations (test and reference formulations) under fasting condition. The AUC was measured based on the plasma concentration of the active metabolite, perindoprilat.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax)of perindopril parent compound | 192 hours
  Relative bioavailability (secondarily measured by Cmax) between two perindopril 4 mg tablet formulations (test and reference formulations) under fasting condition. The Cmax was measured based on the plasma concentration of perindopril parent compound.
Peak plasma concentration (Cmax)of perindoprilat | 192 hours
  Relative bioavailability (secondarily measured by Cmax) between two perindopril 4 mg tablet formulations (test and reference formulations) under fasting condition. The Cmax was measured based on the plasma concentration of the active metabolite, perindoprilat.
Time to achieve the peak plasma concentration (tmax)of perindopril parent compound | 192 hours
Time to achieve the peak plasma concentration (tmax)of perindoprilat | 192 hours
Elimination half-life (t1/2)of perindopril parent compound | 192 hours
Elimination half-life (t1/2)of perindoprilat | 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Danang A Yunaidi, MD, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Bellissant E, Giudicelli JF. Pharmacokinetic-pharmacodynamic model for perindoprilat regional haemodynamic effects in healthy volunteers and in congestive heart failure patients. Br J Clin Pharmacol. 2001 Jul;52(1):25-33. doi: 10.1046/j.0306-5251.2001.01410.x. PMID 11453887
- [Background] Louis WJ, Workman BS, Conway EL, Worland P, Rowley K, Drummer O, McNeil JJ, Harris G, Jarrott B. Single-dose and steady-state pharmacokinetics and pharmacodynamics of perindopril in hypertensive subjects. J Cardiovasc Pharmacol. 1992 Sep;20(3):505-11. doi: 10.1097/00005344-199209000-00024. PMID 1279299
- [Background] Sennesael J, Ali A, Sweny P, Vandenburg M, Slovic D, Dratwa M, Resplandy G, Genissel P, Desche P. The pharmacokinetics of perindopril and its effects on serum angiotensin converting enzyme activity in hypertensive patients with chronic renal failure. Br J Clin Pharmacol. 1992 Jan;33(1):93-9. doi: 10.1111/j.1365-2125.1992.tb04006.x. PMID 1311597